CLINICAL TRIAL: NCT01806350
Title: A Pilot Randomized Control Trial to Evaluate Pelvic Floor Muscle Training for Urinary Incontinence Among Gynecologic Cancer Survivors
Brief Title: Pelvic Floor Muscle Training in Treating Urinary Incontinence in Gynecologic Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: INST 0912; NCI-2012-01319 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-03-05; First posted 2013-03-07 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Cervical Cancer; Endometrial Cancer; Ovarian Epithelial Cancer; Ovarian Germ Cell Tumor; Uterine Sarcoma; Vulvar Cancer
Keywords: Pelvic floor muscle training; incontinence; quality of life
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Carcinoma, Ovarian Epithelial; Vulvar Neoplasms | interventions — Early Intervention, Educational; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (PFMT) (Experimental): Patients receive a handout describing behavioral management tips for urinary incontinence, including information and suggestions about optimal volume fluid intake, constipation management, measures to reduce urgency by spreading fluid intake, and avoiding caffeine and other bladder irritants that have proved effective in other intervention trials. Patients undergo PFMT over 20-30 minutes teaching them to contract the pelvic floor muscles correctly and receive feedback to avoid the contraction of abdominal, gluteal or adductor muscles. Patients are asked to perform 3 sets of 10 pelvic muscle contractions with a goal of holding the contraction for 5 seconds daily for 12 weeks and also receive a reminder phone call to address concerns and review the instructions at 4 weeks.
  Interventions: Other: questionnaire administration; Other: educational intervention
- Arm II (usual care) (Active Comparator): Patients receive usual care for urinary incontinence, with an option to join the training program after completion of study.
  Interventions: Other: questionnaire administration; Procedure: standard follow-up care

INTERVENTIONS:
Other: questionnaire administration — Ancillary studies
Procedure: standard follow-up care — Receive usual care
  Arms: Arm II (usual care)
Other: educational intervention — Undergo PFMT
  Other Names: intervention, educational
  Arms: Arm I (PFMT)

SUMMARY:
This randomized pilot clinical trial studies pelvic floor muscle training in treating urinary incontinence in gynecologic cancer survivors. Pelvic floor muscle training may help control symptoms and improve physical function and quality of life in gynecologic cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether pelvic floor muscle training and behavioral therapy in gynecologic cancer survivors results in improvement in incontinence symptoms as measured by a validated questionnaire (Patient Global Impression of Improvement) at three month follow-up when compared to women who do not undergo pelvic floor muscle training.

II. To evaluate whether women who undergo pelvic floor muscle training and behavioral therapy report greater improvement in validated urinary incontinence symptom severity, pelvic floor distress and quality of life measures than women who do not undergo pelvic floor muscle training.

III. To evaluate the acceptability of pelvic floor muscle training (PFMT) among gynecological cancer survivors and to provide preliminary data to inform a power analysis for a larger randomized trial.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive a handout describing behavioral management tips for urinary incontinence, including information and suggestions about optimal volume fluid intake, constipation management, measures to reduce urgency by spreading fluid intake, and avoiding caffeine and other bladder irritants that have proved effective in other intervention trials. Patients undergo PFMT over 20-30 minutes teaching them to contract the pelvic floor muscles correctly and receive feedback to avoid the contraction of abdominal, gluteal or adductor muscles. Patients are asked to perform 3 sets of 10 pelvic muscle contractions with a goal of holding the contraction for 5 seconds daily for 12 weeks and also receive a reminder phone call to address concerns and review the instructions at 4 weeks.

ARM II: Patients receive usual care for urinary incontinence, with an option to join the training program after completion of study.

After completion of study treatment, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* History of uterine, cervical, ovarian or vulvar malignancy
* Treatment free interval of >= one year and currently have no evidence of cancer
* Reports urinary incontinence based on screening questionnaire
* Must have a stable address for the three month period

Exclusion Criteria:

* Current clinical evidence of urinary tract infection
* Within three months of failed surgery for urinary incontinence
* Planned surgery for urinary incontinence in the next three months
* Presence of neurologic condition that may impact bladder symptoms such as multiple sclerosis, stroke
* Pregnancy

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Improvement in the Patient Global Impression of Improvement (PGI-I) rating | 12 weeks
  Fisher's exact test will be used to test whether the chance of success is identical for the two groups (intervention vs. control).

SECONDARY OUTCOMES:
Changes in the Incontinence Severity Index (ISI) score | Baseline to 3 months
  The Brinks scale will be used by the trainers for the treatment group follow-up to evaluate the adequacy of the contractions in a qualitative manner. A two sample t-test on the within individual differences will be used. A non-parametric Mann-Whitney test will be used if the sample differences are non-normally distributed.
Changes in Urinary Distress Inventory (UDI) | Baseline to 3 months
  The Brinks scale will be used by the trainers for the treatment group follow-up to evaluate the adequacy of the contractions in a qualitative manner. A two sample t-test on the within individual differences will be used. A non-parametric Mann-Whitney test will be used if the sample differences are non-normally distributed.
Changes in Incontinence Impact Questionnaire (IIQ), which measures the impact of urinary incontinence on quality of life | Baseline to 3 months
  The Brinks scale will be used by the trainers for the treatment group follow-up to evaluate the adequacy of the contractions in a qualitative manner. A two sample t-test on the within individual differences will be used. A non-parametric Mann-Whitney test will be used if the sample differences are non-normally distributed.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Rutledge, MD, Principal Investigator — University of New Mexico Cancer Center
Locations (1):
- University of New Mexico Cancer Center, Albuquerque, New Mexico, United States

REFERENCES:
- See also: University of New Mexico Cancer Center — http://www.cancer.unm.edu
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org